CLINICAL TRIAL: NCT07214441
Title: Evaluating the Feasibility and Preliminary Effects of a Remotely Delivered Dyad-Based Intervention Incorporating Resistance Training to Improve Fitness in Individuals With Non-Small-Cell Lung Cancer and in Their Partners
Brief Title: Evaluating the Feasibility and Preliminary Effects of BE+
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Amanda Dyer, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00144866
Record Dates: First submitted 2025-09-12; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer (Non-Small Cell); Self-management Behavior; Physical Activity; Stress; Quality of Life; Resistance Training
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathe Easier+ (Experimental): Breathe Easier+ includes guided instruction using a digital manual, a walking program, RT training sessions, a weekly telephone coaching call, daily text messages, and assessments at three time points.
  Interventions: Behavioral: Breathe Easier+

INTERVENTIONS:
Behavioral: Breathe Easier+ — Breathe Easier+ includes guided instruction using a digital manual, a walking program, RT training sessions, a weekly telephone coaching call, daily text messages, and assessments at three time points.

SUMMARY:
This non-randomized, single group study will test a 12-week, behavioral intervention for physical activity and stress management for survivors of non-small cell lung cancer (NSCLC) and a partner (family member or friend). The goals of this intervention, Breathe Easier+ (BE+), are to increase overall physical activity and overall fitness and to reduce symptoms (fatigue, breathlessness, sleep, and stress).

The aim of this study is to evaluate the enrollment, retention, adherence, participation, and acceptability of the 12-week BE+ among NSCLC survivors and their partners. The study also aims to:

1. Explore preliminary intervention effects of BE+ on increasing physical activity and overall fitness (measured by 7-day Fitbit wear, step-in-place test, chair sit-and-stand, arm curl test, and balance test) from baseline to post-intervention among NSCLC survivors and their partners.
2. Explore preliminary effects of BE+ for improvement in stress response, symptom burden (fatigue, dyspnea), sleep, and HRQL from baseline to post-intervention among NSCLC survivors and their partners.

Participants will receive education, social support, coaching, a guided walking program, supervised resistance training (RT), and meditations delivered via digital technology (tablet, smartphone, and Fitbit).

DETAILED DESCRIPTION:
Lung cancer is the second-most diagnosed malignancy, accounting for more annual deaths than breast, prostate, and colorectal cancers combined. Approximately 80% of lung cancer diagnoses are non-small-cell lung cancer (NSCLC), 42% will present with localized disease and 58% will present with advanced disease. Scientific advances have led to improved 5-year survival rates. These advances are projected to improve, meaning that survivors of NSCLC will live longer. However, the extent of thoracic resection, radiation, chemotherapy, and immunotherapy treatment; common comorbid conditions like COPD (chronic obstructive pulmonary disease); and health behaviors exacerbate physical and emotional health burdens. Research has yet to address the management of physical deconditioning and unresolved symptoms (e.g., dyspnea, fatigue) in long-term survivors of lung cancer, both of which negatively impact health-related quality of life (HRQL). Self-management interventions that target lifestyle behaviors such as physical activity and stress reduction have demonstrated meaningful benefit in managing symptom burden. Additionally, scientific consensus supports the use of resistance training (RT) to mitigate functional decline from physical deconditioning by increasing muscular strength and endurance. However, frequently NSCLC survivors are sedentary or insufficiently active.

Lifestyle behaviors tend to cluster in families and social networks; thus, family members and friends of survivors are also at risk of poor health. An emerging consensus corroborates the inclusion of family and friends ("partners") of cancer survivors in self-management interventions. In this proposal, a partner is anyone the survivor considers a supportive person. Partners are critical sources of all types of social support across the cancer continuum. Importantly, partners must cope with their own concerns, including uncertainty surrounding the survivor's illness, fear of losing their partner, and the impact of their own health behaviors. Together, survivors and their partners may benefit significantly from a dyad-based lifestyle behavior intervention that supports physical and emotional health.

This research team has conducted extensive formative and preliminary research to develop a dyad-based intervention for NSCLC survivors and their partners. Early on, participants clearly indicated a preference for home-based, family- and safety-oriented interventions. Most recently, participants demonstrated the feasibility and preliminary effectiveness of a 12-week, dyad-based, telephone-delivered, self-management intervention known as Breathe Easier (BE), featuring mindfulness-based breathing exercises, meditation, and a walking program for dyads (N = 40; 20 dyads). Another study involved testing an RT program tailored to survivors only (n = 14). Feasibility and acceptability were strong and indicated positive improvements involving symptom burden and physical functioning.

Recognizing that evidence supports a multimodal approach, our research team aims to expand the BE intervention by integrating home-based RT via digital technology. The revised intervention will be known as BE+ and will include stage IV survivors to better understand the feasibility of this subgroup.

Theoretical Approach: The ORBIT model, which is a systematic framework for developing behavioral interventions, was used to develop a chain of evidence for the BE+ intervention program. BE+ is also built on the individual and family self-management theory (IFSMT), which proposes that successful change in health behavior self-management after a diagnosis of lung cancer requires active involvement by the survivor coupled with partner support. IFSMT encompasses three broad dimensions (context, process, outcomes) and promotes self-regulation, self-efficacy, and social support. The context dimension may impact individual and partner engagement in the self-management process and, therefore, the outcomes. Within the process dimension, self-regulation of the self-management of behaviors requires active involvement. Social support enhances the capacity to change and influences collaboration among dyads. The program components of BE+ enhance these three factors-leading to improved health behaviors. The behaviors of individuals in close, personal relationships are interdependent, and the actions of one person continuously affect the other's actions.

Design: A 12-week, non-randomized, one group pre-post feasibility study piloted among NSCLC survivors and their partners.

A purposive sample of 10 dyads (N = 20 participants) will be recruited from two cancer treatment centers in South Carolina. A partner, defined as a relative or close friend (i.e., spouse, sibling, adult child, neighbor), will be required for enrollment.

Analysis Plan: A power analysis will not be performed as this feasibility study does not warrant formal hypothesis testing, and all statistical tests will use an α cut point of 0.10 for meaningful preliminary differences. This nontraditional cut point (vs. α = 0.05) is more lenient due to the feasibility study design. Data analysis software will be used to obtain information regarding step count, and sleep SAS 9.4 (Cary, NC) software will be used to calculate means (± SD) and frequencies for demographic data. Normality will be checked using histogram and Q-Q plots combined with skewness and kurtosis statistics. When the outcome is normally distributed, independent t-tests will be performed to assess subset differences between survivors and partners to evaluate preliminary effects. Equal variances will be determined using the Folded F test, and thus the pooled version of the independent t-test will be used to determine preliminary meaningful differences. Then repeated measures ANOVA will be used to compare means among three time points. If normality is violated, the Mann-Whitney U Test will be used to compare outcome differences between survivors and partners, and Friedman's ANOVA by ranks will be used to evaluate the differences among three time points.

Exit interviews will be audio-recorded and professionally transcribed. The lead investigator will review transcripts and audio recordings to confirm accuracy. Thematic analysis will be used to analyze the transcripts following a six-phase approach: (1) become familiar with the data, (2) generate codes, (3) search for themes, (4) review themes, (5) define or name themes, (6) report findings and analysis.64 Transcripts will be iteratively analyzed by the research team to reach a consensus on codes, categories, and themes.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of NSCLC who have completed definitive treatment within the last 2 years.
* All participants must have a health clearance for physical activity signed by a healthcare provider; have Wi-Fi access; be able to provide informed consent; and be able to speak and read English.

Exclusion Criteria:

* Survivors on current definitive treatment.
* All participants with a history of recurrent falls; a substantial mobility impairment related to chronic disease or injury; and lack of physical activity readiness as determined by a healthcare provider.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of the 12-week BE+ (BE with RT) among NSCLC survivors and their partners (dyads). | 12 weeks
  Feasibility will be evaluated on:
  1. Enrollment (25% of eligible participants),
  2. Retention (80% of participants at study completion),
  3. Adherence (80% to complete instruments at time points 1-3; Fitbit wear >5 days each week for 12 weeks),
  4. Participation (80% to log physical activity weekly, log breathing exercises weekly, set goals weekly, attend 2 resistance training sessions weekly, participate in weekly phone call, and read daily text messages),

SECONDARY OUTCOMES:
Explore preliminary effects of BE+ on increasing physical activity and overall fitness from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  Physical activity and overall fitness will be measured:
  7-Day Fitbit Step Count: 7-day total steps, measured during activity tracking, including active zone minutes and step counting for 24 hours/day, found to be accurate with an absolute percent error for steps of 1.5-9.6%.
  Sit-to-Stand Test: Evaluates how long a person takes to rise from a chair and return to sitting in the chair, 5 times consecutively. Measured in seconds. A reliable and widely accepted measure of physical function. ICC = 0.937.
  Step-in-Place Test: 2-minute marching in place, to estimate aerobic endurance; score is the number of times the right knee reaches the target, which has been validated with ICC = 0.90, correlation coefficient (r) = 0.69.
  Arm Curl Test: 30 seconds of arm curls holding a weight to measure upper body strength and muscular endurance; ICC = 0.88.
  Single Leg Stance: Length of time participant can stand on 1 leg with hands on hips to limit movement of arms; ICC = 0.87-0.97.
Explore preliminary effects of BE+ for reduction in dyspnea from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  mMRC Dyspnea Scale: 1 item correlates with a self-report of breathlessness. Sensitivity (0.21-0.68), specificity (0.91-1.0).
Explore preliminary effects of BE+ for reduction in stress response from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  Fitbit Heart Rate Variability (HRV): Measure of the fluctuation of the length of heartbeat intervals, representing the ability of the heart to respond to varying physiological stimuli, signifying stress response. ICC = 0.6
Explore preliminary effects of BE+ for improvement in sleep from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  Fitbit Sleep: Objective measure of sleep quantity based on combined body movement and HRV algorithm. Sleep measures captured by Fitbit include total minutes asleep, minutes awake, minutes to fall asleep, minutes awake after sleep, total time in bed, and sleep stages. Sensitivity = .95; specificity = 0.58-0.69.
  Pittsburgh Sleep Quality Index (PSQI): 19 items measuring sleep quality, sleep latency, sleep efficiency, sleep duration, sleep disturbances, use of sleep medications, and daytime dysfunction.55 Cronbach's alpha (α) = 0.77-0.83; r = 0.77-0.85.
Explore preliminary effects of BE+ for reduction in fatigue from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  FACIT Fatigue Scale v.4: 13 items measuring fatigue during usual activity over the past 7 days. α = 0.96; ICC = 0.95.
Explore preliminary effects of BE+ for improvement in health-related quality of life (HRQL) from baseline to post-intervention among NSCLC survivors and their partners (dyads). | 12 weeks
  Short Form Health Survey (SF-36): 36 items evaluating HRQL through physical function, social functioning, physical role limitations, emotional role limitations, emotional health, vitality, pain, and general health perception. α = 0.78-0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Lee EC, Whitehead AL, Jacques RM, Julious SA. The statistical interpretation of pilot trials: should significance thresholds be reconsidered? BMC Med Res Methodol. 2014 Mar 20;14:41. doi: 10.1186/1471-2288-14-41. PMID 24650044
- [Background] Beck SL, Schwartz AL, Towsley G, Dudley W, Barsevick A. Psychometric evaluation of the Pittsburgh Sleep Quality Index in cancer patients. J Pain Symptom Manage. 2004 Feb;27(2):140-8. doi: 10.1016/j.jpainsymman.2003.12.002. PMID 15157038
- [Background] Dorn LD, Lucke JF, Loucks TL, Berga SL. Salivary cortisol reflects serum cortisol: analysis of circadian profiles. Ann Clin Biochem. 2007 May;44(Pt 3):281-4. doi: 10.1258/000456307780480954. PMID 17456296
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Tsiligianni IG, Alma HJ, de Jong C, Jelusic D, Wittmann M, Schuler M, Schultz K, Kollen BJ, van der Molen T, Kocks JW. Investigating sensitivity, specificity, and area under the curve of the Clinical COPD Questionnaire, COPD Assessment Test, and Modified Medical Research Council scale according to GOLD using St George's Respiratory Questionnaire cutoff 25 (and 20) as reference. Int J Chron Obstruct Pulmon Dis. 2016 May 18;11:1045-52. doi: 10.2147/COPD.S99793. eCollection 2016. PMID 27274226
- [Background] Ponce-Gonzalez JG, Sanchis-Moysi J, Gonzalez-Henriquez JJ, Arteaga-Ortiz R, Calbet JA, Dorado C. A reliable unipedal stance test for the assessment of balance using a force platform. J Sports Med Phys Fitness. 2014 Feb;54(1):108-17. PMID 24445552
- [Background] Melo TA, Duarte ACM, Bezerra TS, Franca F, Soares NS, Brito D. The Five Times Sit-to-Stand Test: safety and reliability with older intensive care unit patients at discharge. Rev Bras Ter Intensiva. 2019;31(1):27-33. doi: 10.5935/0103-507X.20190006. Epub 2019 Mar 14. PMID 30892478
- [Background] Chen MD, Kuo CC, Pellegrini CA, Hsu MJ. Accuracy of Wristband Activity Monitors during Ambulation and Activities. Med Sci Sports Exerc. 2016 Oct;48(10):1942-9. doi: 10.1249/MSS.0000000000000984. PMID 27183123
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Kim M, Yeom HE, Jung MS. Validation and psychometric properties of the multidimensional scale of perceived social support among Korean breast cancer survivors. Asia Pac J Oncol Nurs. 2022 Jan 30;9(4):229-235. doi: 10.1016/j.apjon.2022.01.004. eCollection 2022 Apr. PMID 35571625
- [Background] McDonnell KK, Gallerani DG, Newsome BR, Owens OL, Beer J, Myren-Bennett AR, Regan E, Hardin JW, Webb LA. A Prospective Pilot Study Evaluating Feasibility and Preliminary Effects of Breathe Easier: A Mindfulness-based Intervention for Survivors of Lung Cancer and Their Family Members (Dyads). Integr Cancer Ther. 2020 Jan-Dec;19:1534735420969829. doi: 10.1177/1534735420969829. PMID 33118443
- [Background] Cooley ME, Blonquist TM, Hong F, Nayak MM, Crouter SE, Hayman LL, Jaklitsch MT, Emmons KM, Bueno R. The effect of a lifestyle risk reduction intervention on lifestyle adherence and health-related quality of life in nonsmall cell lung cancer survivors: Feasibility study outcomes. Psychooncology. 2019 Apr;28(4):920-923. doi: 10.1002/pon.5002. Epub 2019 Feb 12. No abstract available. PMID 30673155
- [Background] Blok AC, Blonquist TM, Nayak MM, Somayaji D, Crouter SE, Hayman LL, Colson YL, Bueno R, Emmons KM, Cooley ME. Feasibility and acceptability of "healthy directions" a lifestyle intervention for adults with lung cancer. Psychooncology. 2018 Jan;27(1):250-257. doi: 10.1002/pon.4443. Epub 2017 May 31. PMID 28426922
- [Background] Heredia-Ciuro A, Martin-Nunez J, Lopez-Lopez JA, Lopez-Lopez L, Granados-Santiago M, Calvache-Mateo A, Valenza MC. Effectiveness of healthy lifestyle-based interventions in lung cancer survivors: a systematic review and meta-analysis. Support Care Cancer. 2022 Dec 21;31(1):71. doi: 10.1007/s00520-022-07542-0. PMID 36542189
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Roddy MK, Flores RM, Burt B, Badr H. Lifestyle behaviors and intervention preferences of early-stage lung cancer survivors and their family caregivers. Support Care Cancer. 2021 Mar;29(3):1465-1475. doi: 10.1007/s00520-020-05632-5. Epub 2020 Jul 20. PMID 32691229
- [Background] Nightingale CL, Steffen LE, Tooze JA, Petty W, Danhauer SC, Badr H, Weaver KE. Lung Cancer Patient and Caregiver Health Vulnerabilities and Interest in Health Promotion Interventions: An Exploratory Study. Glob Adv Health Med. 2019 Jul 17;8:2164956119865160. doi: 10.1177/2164956119865160. eCollection 2019. PMID 31360617
- [Background] McDonnell KK, Owens OL, Hilfinger Messias DK, Heiney SP, Friedman DB, Campbell C, Webb LA. Health behavior changes in African American family members facing lung cancer: Tensions and compromises. Eur J Oncol Nurs. 2019 Feb;38:57-64. doi: 10.1016/j.ejon.2018.12.002. Epub 2018 Dec 7. PMID 30717937
- [Background] Cooley ME, Finn KT, Wang Q, Roper K, Morones S, Shi L, Litrownik D, Marcoux JP, Zaner K, Hayman LL. Health behaviors, readiness to change, and interest in health promotion programs among smokers with lung cancer and their family members: a pilot study. Cancer Nurs. 2013 Mar-Apr;36(2):145-54. doi: 10.1097/NCC.0b013e31825e4359. PMID 22791213
- [Background] Sande-Rivadulla M, Alonso-Calvete A, Soto-Gonzalez M. Effects of Muscle Strength Training in Prostate Cancer: A Systematic Review. Arch Esp Urol. 2024 Jan;77(1):1-15. doi: 10.56434/j.arch.esp.urol.20247701.1. PMID 38374007
- [Background] Chodosh J, Morton SC, Mojica W, Maglione M, Suttorp MJ, Hilton L, Rhodes S, Shekelle P. Meta-analysis: chronic disease self-management programs for older adults. Ann Intern Med. 2005 Sep 20;143(6):427-38. doi: 10.7326/0003-4819-143-6-200509200-00007. PMID 16172441
- [Background] Vijayvergia N, Shah PC, Denlinger CS. Survivorship in Non-Small Cell Lung Cancer: Challenges Faced and Steps Forward. J Natl Compr Canc Netw. 2015 Sep;13(9):1151-61. doi: 10.6004/jnccn.2015.0140. PMID 26358799
- [Background] Newsome BR, McDonnell K, Hucks J, Dawson Estrada R. Chronic Obstructive Pulmonary Disease: Clinical Implications for Patients With Lung Cancer. Clin J Oncol Nurs. 2018 Apr 1;22(2):184-192. doi: 10.1188/18.CJON.184-192. PMID 29547609
- [Background] Lowery AE, Krebs P, Coups EJ, Feinstein MB, Burkhalter JE, Park BJ, Ostroff JS. Impact of symptom burden in post-surgical non-small cell lung cancer survivors. Support Care Cancer. 2014 Jan;22(1):173-80. doi: 10.1007/s00520-013-1968-3. Epub 2013 Sep 10. PMID 24018910
- [Background] Granger CL, McDonald CF, Irving L, Clark RA, Gough K, Murnane A, Mileshkin L, Krishnasamy M, Denehy L. Low physical activity levels and functional decline in individuals with lung cancer. Lung Cancer. 2014 Feb;83(2):292-9. doi: 10.1016/j.lungcan.2013.11.014. Epub 2013 Nov 26. PMID 24360323
- [Background] Miller KD, Nogueira L, Devasia T, Mariotto AB, Yabroff KR, Jemal A, Kramer J, Siegel RL. Cancer treatment and survivorship statistics, 2022. CA Cancer J Clin. 2022 Sep;72(5):409-436. doi: 10.3322/caac.21731. Epub 2022 Jun 23. PMID 35736631
- [Background] McDonnell KK, Estrada RD, Dievendorf AC, Blew L, Sercy E, Khan S, Hardin JW, Warden D, Eberth JM. Lung cancer screening: Practice guidelines and insurance coverage are not enough. J Am Assoc Nurse Pract. 2019 Jan;31(1):33-45. doi: 10.1097/JXX.0000000000000096. PMID 30431549
- See also: American Cancer Society. (2025). Cancer facts and figures 2025. — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/2025-cancer-facts-figures.html